CLINICAL TRIAL: NCT07398170
Title: Search for Circulating Tumour Cells in the Blood and/or Cerebrospinal Fluid in Patients With Recurrent Aggressive Meningiomas That Have Recurred: Proof-of-concept Study
Brief Title: Search for Circulating Tumour Cells in the Blood and/or Cerebrospinal Fluid in Patients With Recurrent Aggressive Meningiomas: Proof-of-concept Study
Acronym: BIOLIMEN-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL24_0381
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Meningioma
Keywords: Meningioma diagnosis; Circulating tumor cells; Liquid Biopsy; Neoplasm Recurrence, Local; Therapy; Biomarkers
MeSH Terms: conditions — Meningioma; Neoplastic Cells, Circulating; Neoplasm Recurrence, Local | interventions — Blood Specimen Collection; Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental)
  Interventions: Other: Blood sampling; Other: Lumbar puncture

INTERVENTIONS:
Other: Blood sampling — At the diagnosis of meningioma recurrence: a blood sample of 28 mL of whole blood (i.e., 4 EDTA tubes of 7 mL each) and at the end of meningioma recurrence treatment: a blood sample of 28 mL of whole blood (i.e., 4 EDTA tubes of 7 mL each) will be collect.
Other: Lumbar puncture — At the time of diagnosis of meningioma recurrence :a cerebrospinal fluid (CSF) sample obtained by lumbar puncture, in the absence of contraindications verified by the investigator, collected in one dry tube of 4 mL.

SUMMARY:
The goal of the clinical trial is to assess the presence of circulating tumor cells (CTCs) in the blood and/or cerebrospinal fluid (CSF) of patients with aggressive recurrent meningiomas.

DETAILED DESCRIPTION:
Meningiomas are the most common intracranial tumours. In 80% of cases, they are benign (grade I) and have an indolent growth profile. These tumours are monitored radiologically and clinically using magnetic resonance imaging (MRI), or treated by surgical excision, with good results. However, 20% of them manifest as more aggressive tumours, leading to significant morbidity, either due to symptoms related to their natural history or complications related to treatment. These aggressive meningiomas represent a challenge both in terms of prognosis assessment and treatment selection.

Meningiomas are generally diagnosed using a CT or MRI scan of the brain or spinal cord with contrast injection. However, a definitive diagnosis remains dependent on histopathology, which is used to decide on the treatment sequence.

Recently, liquid biopsy has proven useful in the diagnosis and monitoring of many cancerous conditions. However, no studies have been conducted on the presence of circulating tumour cells (CTCs) in meningiomas. Although these tumours are intracranial, they develop outside the blood-brain barrier, so it is likely that cells are detectable in the blood and cerebrospinal fluid (CSF).

The use of blood markers could enable non-invasive confirmation of the diagnosis when a meningioma is detected by imaging, as well as assessment of the risk of recurrence in the post-operative period.

The BIOLIMEN-1 study is a pilot study aimed at developing and validating this concept.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Operated on for a grade 2 or 3 meningioma at Montpellier University Hospital between 2015 and 2024
* Tumour expressing SSTR2A on the initial surgical specimen
* Clinical and/or radiological recurrence as determined by MRI imaging (progression of a residual lesion OR appearance of a new lesion consistent with a meningioma at the surgical site or elsewhere)

Exclusion Criteria:

* Other active ongoing cancer
* Contraindications to lumbar puncture:
* Intracranial hypertension with meningioma exerting a mass effect and obstruction of the cerebrospinal fluid (CSF) pathway/risk of trans-tentorial or amygdalar herniation
* Blood clotting disorder with risk of haematoma at the puncture site (anticoagulant treatment at therapeutic dose or antiplatelet therapy, thrombocytopenia or thrombopathy)
* Infection at the puncture site
* Pregnant or breastfeeding women (Article L.1121-5 of the French Public Health Code)
* Persons deprived of their liberty by judicial or administrative decision (Article L.1121-6 of the French Public Health Code)
* Persons who are subject to legal protection measures or who are unable to express their consent (guardianship, curatorship, judicial protection; Article L.1121-8 of the French Public Health Code)
* Not affiliated with a social security scheme or beneficiary of such a scheme (Article L.1121-8-1 of the French Public Health Code)
* Persons participating in another study that includes an ongoing exclusion period (Article L.1121-12 of the French Public Health Code)
* Failure to obtain written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Detection rate of circulating tumour cells (CTC) in blood | Before treatment of meningioma recurrence and at the end of meningioma recurrence treatment on Day 90 (± 15 days) in case of radiotherapy, or on Day 1 post-surgery in case of surgery
  i.e the proportion of patients with at least one CTC in the venous blood sample
Detection rate of circulating tumour cells (CTC) in cerebrospinal fluid | Before treatment of meningioma recurrence
  i.e the proportion of patients with at least one CTC in the cerebrospinal fluid

SECONDARY OUTCOMES:
Presence of circulating tumour cells (CTC) in blood | Before treatment of meningioma recurrence and at the end of meningioma recurrence treatment on Day 90 (± 15 days) in case of radiotherapy, or on Day 1 post-surgery in case of surgery
  i.e defined as the presence of at least one CTC in the blood sample
Presence of circulating tumour cells (CTC) in cerebrospinal fluid | Before treatment of meningioma recurrence
  i.e defined as the presence of at least one CTC in the cerebrospinal fluid sample
Number of circulating tumour cells (CTC) in blood | Before treatment of meningioma recurrence and at the end of meningioma recurrence treatment on Day 90 (± 15 days) in case of radiotherapy, or on Day 1 post-surgery in case of surgery
Number of circulating tumour cells (CTC) in cerebrospinal fluid | Before treatment of meningioma recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Montpellier, Montpellier, France, France

IPD SHARING:
Plan to Share IPD: Undecided